CLINICAL TRIAL: NCT03046862
Title: Biomarker-oriented Study of Durvalumab(MEDI4736)/Tremelimumab in Combination With Gemcitabine/Cisplatin in Chemotherapy-naïve Biliary Tract Cancer
Brief Title: Durvalumab(MEDI4736)/Tremelimumab in Combination With Gemcitabine/Cisplatin in Chemotherapy-naïve Biliary Tract Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Do-Youn Oh, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTC-1st MEDITREME
Record Dates: First submitted 2017-02-06; First posted 2017-02-08 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Biliary Tract Neoplasms
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — durvalumab; tremelimumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Durvalumab/Tremelimumab+chemotherapy (Experimental): Durvalumab and Tremelimumab in combination with gemcitabine/cisplatin.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Durvalumab — Durvalumab 1.12 g iv on D1 every 3 weeks
  Other Names: MEDI4736
Drug: Tremelimumab — Tremelimumab 75mg iv on D1 every 3 weeks
Drug: Gemcitabine — Gemcitabine 1000 mg/m2 iv on D1& D8 every 3 weeks
Drug: Cisplatin — Cisplatin 25 mg/m2 iv on D1& D8 every 3 weeks

SUMMARY:
<Research Hypothesis> The dynamics of immune systems by cytotoxic chemotherapy and its changes by combination with immuno-oncology agents will be uncovered.

The combination of Durvalumab/Tremelimumab with gemcitabine/cisplatin chemotherapy is feasible and efficacious in chemo-naïve biliary tract cancer.

<Purpose of the study> To assess the effect of Durvalumab/Tremelimumab in combination with gemcitabine/cisplatin on response rate (RR) in chemo-naïve advanced biliary tract cancer patients.

DETAILED DESCRIPTION:
<Rationale for conducting this study>

1. Rational #1. The incidence of biliary tract cancer (BTC) is higher in Korea than the West. (Korea: 10 new cases/100,000 population every year, the West:1-2 cases/100,100 population every year). Therefore, to conduct clinical study of BTC in Korea is very feasible and efficient.
2. Rational #2 The Gemcitabine/cisplatin is the current standard of care in 1st-line treatment for advanced BTC ((N Engl J Med 2010; 362 (14): 1273-81). No one-targeted therapy has been approved in BTC, yet. The overall survival of advanced BTC with cytotoxic chemotherapy is only 8-10 months, in general. Therefore, there is a huge unmet medical need.
3. Rational #3 In recent sequencing data of BTC showed the BTC patients with the worse prognosis had significant enrichment of hypermutated tumors and a characteristic elevation in the expression of immune checkpoint molecules. According, immune-modulating therapies also be potentially promising options for these patients (Nat Genet. 2015 Sep;47(9):1003-10.)
4. Rational #4 In PDL1 (+) BTC, anti-PD1 Ab shows promising activity as a monotherapy (Bang YJ, et al. ECC/ESMO 2015) In one clinical study of pembrolizumab, 37 out of 89 BTC patients (41.6%) showed the PDL1 (+) tumor. Among 24 PDL1 (+) patients who were enrolled and treated with pembrolizumab, 50% were Asian, 62.5% had ECOG 1, 16.7% had gallbladder cancer, 80% were at the 3rd-line or later setting. Four patients showed PR (3 from Seoul National University Hospital), 4 patients SD, which led the overall response rate of 17.4%. A total 40% of patients showed tumor shrinkage. The decreases in tumor size were generally maintained over time. This study gives us the evidence that immune checkpoint inhibitor is working on BTC likewise other solid tumors.
5. Rational #5 In recent studies have shown the combination of CTLA4 inhibitor with anti-PD1/PDL1 agents shows the enhanced clinical activities, especially, regardless of PDL1 status. This combination strategy is being actively under test in many solid tumors.
6. Rational #6 Certain chemotherapeutic drugs stimulate cancer-specific immune responses by inducing immunogenic cell death and other effector mechanisms (Immunity 2013, Annu Rev Immunol 2013) With the cytotoxic chemotherapy, the PDL-1 is induced and this increased expression of PDL1 contributes the resistance to cytotoxic chemotherapy. Successful eradication of tumors by immunogenic chemotherapy requires removal of immunosuppressive IgA+, PDL1+plasmocytes (Nature 2015). More importantly, still vast majorities of dynamic changes of immune system by cytotoxic chemotherapy are unanswered.

   These support that the combination of cytotoxic chemotherapy with immuno-oncology agents including immune checkpoint inhibitors might be efficacious and needed.
7. Rational #7 The advantages of "Immunotherapy and cytotoxic chemotherapy" combination are; 1) can explore science on the dynamic immunologic changes by cytotoxic chemotherapy and its overcome by immunotherapy 2) easy way to be incorporated in the current clinical practice 3) can be applied to variety of tumor types such as NSCLC, urothelial cancer. 4) relatively affordable than "immunotherapy and targeted agent" combination. Durvalumab/Tremelimumab in combination of cytotoxic chemotherapy has not been tested, especially in BTC.

<Sample Size Determination> Primary efficacy endpoint is response rate. In BTC, the response rate of 1st-line gemcitabine/cisplatin chemotherapy is about 20% (20% in BT22 clinical trial, 25% in ABC-02 clinical trial). Therefore, we set H0 as 20%, and H1 as 40%. Using 75% of power and a-error of 0.05, a total 28 patients will be needed. When we assume the drop-out rate of 10%, a total of 31 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven BTC, including intrahepatic cholangiocarcinoma, extrahepatic bile duct cancer, gallbladder cancer, ampulla of vater cancer
* Unresectable or recurrent
* chemotherapy -naïve for their unresectable or recurrent cancer (Previous expose to adjuvant chemotherapy is allowed)
* should have measurable lesion
* ECOG 0, 1
* Without previous expose to immune-oncology agents including anti-CTLA4, anti-PD1, anti-PDL1, etc
* Adequate organ function

  : ANC>1500/mm3, platelet>100K/mm3, HgB>9 g/Dl, bilirubin<1.5 x ULN, ALT/AST<2.5 X UNL, (in case of liver metastasis, <5 Xunl), Cr<1.5 mg/Dl
* Informed consent

Exclusion Criteria:

* Previous treatment for unresectable or recurrent cancer
* Under immunosuppressive agents higher than equivalent dose of prednisone 10mg/day
* Uncontrolled disease such as current active infection, congestive heart failure, uncontrolled hypertension, unstable angina, arrhythmia, interstitial lung disease
* Current active pulmonary tuberculosis
* Current active hepatitis B or hepatitis C (simple carrier is allowed)
* anti-HIV (+)
* Pregnant, breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-02-25 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Response rate | 6 weeks
  According to RECIST v1.1 criteria

SECONDARY OUTCOMES:
Disease control rate | 6 weeks
  the percentage of patients who have achieved complete response, partial response and stable disease
Progression-free survival | 6 weeks
  Time from randomization until disease progression or death
Duration of response | 1 year
  Time from documentation of tumor response to disease progression
Overall survival | 1 year
  Time from randomization until death from any cause
Quality-of-life as measured by EORTC QLQ-BIL21 | 1 year
  EORTC QLQ-BIL21
Overall response rate | 6 week
  According to immune-related response criteria
Safety and tolerability as measured by number and grade of toxicity events | 6 week
  CTCAE V4.1

CONTACTS AND LOCATIONS:
Overall Officials: Do-Youn Oh, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oh DY, Lee KH, Lee DW, Yoon J, Kim TY, Bang JH, Nam AR, Oh KS, Kim JM, Lee Y, Guthrie V, McCoon P, Li W, Wu S, Zhang Q, Rebelatto MC, Kim JW. Gemcitabine and cisplatin plus durvalumab with or without tremelimumab in chemotherapy-naive patients with advanced biliary tract cancer: an open-label, single-centre, phase 2 study. Lancet Gastroenterol Hepatol. 2022 Jun;7(6):522-532. doi: 10.1016/S2468-1253(22)00043-7. Epub 2022 Mar 9. PMID 35278356